CLINICAL TRIAL: NCT01763632
Title: Development of Transcutaneous Bilirubin Nomogram to Identify Neonatal Hyperbilirubinemia in Term and Late-preterm Infants: a Multicenter Study in China
Brief Title: Development of TcB Nomogram to Identify Neonatal Hyperbilirubinemia in Term and Late-preterm Infants
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: Children's Hospital of Fudan University (Other); Nanjing Maternity and Child Health Care Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Jinlin Provincial Maternal and Child Health Hospital (Unknown); Peking University Third Hospital (Other); Inner Mongolia Maternal and Child Health Care Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Guangdong Women and Children Hospital (Other); Guangxi Maternal and Child Health Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Sichuan Provincial People's Hospital (Other); Guiyang Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Principal Investigator, Nanjing Medical University
Other Study IDs: NMU-FY2012-318
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; Neonatal; Transcutaneous Bilirubin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Transcutaneous bilirubinometry — Device: JM-103 (Minolta, Osaka, Japan, jaundice assessment) Procedure: Transcutaneous bilirubinometry (TcB)

SUMMARY:
Thirteen hospitals in China will participate in the study, which aims to provide data on transcutaneous bilirubin (TcB) levels for the first 168 hr after birth in term and late-preterm neonates, and develop an hour-specific TcB nomogram.

The investigators hypothesize that the hour-specific TcB nomogram can predict neonatal hyperbilirubinemia in term and late-preterm Chinese infants, and plan appropriate follow-up for hyperbilirubinemia in newborns.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia is very common; it is not always a benign condition. If left untreated, it can have devastating consequences including cerebral palsy and hearing loss. It is therefore critical to be able to identify the newborns at risk for severe hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

Term or late-preterm newborn infants with GAs of ≥35 weeks and birth weights of ≥2,000 g were included.

Exclusion Criteria:

All sick newborn infants who were admitted to the intensive care unit.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term or late-preterm newborn infants from thirteen hospital in China were recruited.
Sampling Method: Probability Sample
Enrollment: 19601 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change of transcutaneous bilirubin levels from baseline to each postpartum examination up to 168 hr after birth | Every 12 hr for 168 hr.
  During the first postnatal day, transcutaneous bilirubin (TcB) measures were performed at 12-hour time intervals up to the age of 168 hr. TcB data are used to develop an hour-specific TcB nomogram.

SECONDARY OUTCOMES:
Predictive ability of an hour-specific TcB nomogram | At the 28 days after birth
  Evaluate the rate of rise of bilirubin for different time periods and percentile curves and to assess predictive ability of these percentile curves for hyperbilirubinemia, defined as requirement of phototherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chen, PhD, Study Director — Children's Hospital of Fudan University; Shuping Han, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Zhangbin Yu, PhD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital; Chunming Jiang, PhD, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Yan Gao, PhD, Principal Investigator — Jinlin Provincial Maternal and Child Health Hospital; Xiaomei Tong, PhD, Principal Investigator — Peking University Third Hospital; Meihua Pu, PhD, Principal Investigator — Peking University Third Hospital; Hongyun Wang, PhD, Principal Investigator — Inner Mongolia Maternal and Child Health Care Hospital; Kezhan Liu, PhD, Principal Investigator — Shanxi Provincial Maternity and Children's Hospital; Jin Wang, PhD, Principal Investigator — Children's Hospital of Fudan University; Jimei Wang, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University; Xiuyong Cheng, PhD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Jie Yang, PhD, Principal Investigator — Guangdong Women and Children Hospital; Qiufen Wei, PhD, Principal Investigator — Guangxi Maternal and Child Health Hospital; Zhankui Li, PhD, Principal Investigator — Shanxi Provincial Maternity and Children's Hospital; Mingxia Li, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Ling Liu, PhD, Principal Investigator — Guiyang Maternity and Child Health Care Hospital; Xiaofan Sun, MD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital
Locations (15):
- China (15):
  - Guangdong Maternal and Children's Hospital, Guangzhou Medical College, Guangzhou, Guangdong
  - Guangxi Maternal and Child Health Hospital, Liuchow, Guangxi
  - Guiyang Maternal and Child Health Hospital, Guiyang, Guizhou
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Inner Mongolia Maternal and Child Health Care Hospital, Hohhot, Inner Mongolia
  - Nanjing Maternity and Child Health Care Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jinlin Provincial Maternal and Child Health Hospital, Changchun, Jilin
  - Shaanxi Provincial Maternal and Child Health Hospital, Taiyuan, Shaanxi
  - Shaanxi Provincial Maternal and Child Health Hospital, Xi'an, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Third Hospital of Peking University, Beijing
  - Gynecology and Obstetrics Hospital, Fudan University, Shanghai
  - Children's Hospital of Fudan University, Shanghai